CLINICAL TRIAL: NCT07155421
Title: Effects of Early Cardiopulmonary Rehabilitation in Patients With Acute Decompensated Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Saglik Bilimleri Universitesi (Other); Yeditepe University (Other)
Responsible Party: Principal Investigator, Melih Zeren, Associate Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bakircaymzeren09
Record Dates: First submitted 2025-08-25; First posted 2025-09-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early cardiopulmonary rehabilitation group (Experimental): Exercise-based cardiopulmonary rehabilitation will be applied to this group during the hospital stay every day for 3 times a day.
  Interventions: Other: Early Cardiopulmonary Rehabilitation; Other: Routine in-hospital care
- Control Group (Other): Routine in-hospital care will be applied to this group.
  Interventions: Other: Routine in-hospital care

INTERVENTIONS:
Other: Early Cardiopulmonary Rehabilitation — An individualized CPR program including positioning, deep breathing exercises (diaphragmatic and segmental breathing exercises), pursed-lip breathing exercises, breathing exercises using incentive spirometry, and progressive mobilization exercises (in-bed range of motion exercises, sitting, standing, and walking exercises)
  Arms: Early cardiopulmonary rehabilitation group
Other: Routine in-hospital care — Routine in-hospital care for acute decompansated heart failure

SUMMARY:
Acute decompensated heart failure (ADHF) is a severe condition characterized by rapid deterioration of cardiac function, leading to impaired oxygen delivery and multi-organ dysfunction. ADHF often results in reduced physical and respiratory capacity, greater dependence on oxygen support, difficulty performing daily activities, and prolonged hospital stays. In recent years, early exercise-based cardiopulmonary rehabilitation (CPR) has been introduced as part of heart failure management. Evidence suggests that early CPR improves overall health and cardiac function in heart failure patients. However, data regarding its effects in ADHF remain limited. While some studies indicate that early CPR enhances physical function, its impact on respiratory parameters and clinical outcomes is less well established.

Cardiopulmonary rehabilitation is a multidisciplinary program designed to promote physical, psychological, and social recovery in patients with cardiovascular and pulmonary diseases. It includes exercise training, education, psychosocial support, and behavioral strategies. Early CPR specifically aims to improve cardiovascular and respiratory functions in heart failure patients. Initiating CPR in the early phase of ADHF may accelerate recovery, strengthen cardiopulmonary function, shorten hospitalization, and improve quality of life.

This study aims to evaluate the effects of early CPR on functional capacity, hemodynamic parameters, and respiratory parameters in patients with ADHF.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with a diagnosis of acute decompensated heart failure
* Being clinically stable

Exclusion Criteria:

* Having diagnosed pulmonary, neurological, renal, liver, gastrointestinal, orthopedic or oncological pathologies
* Having cardiomyopathy or congestive pericarditis
* Recent heart surgery in the past 6 months
* New or suspected thromboembolic event
* Presence of open wounds, ulcerations or major dermatological diseases in the lower extremities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | At baseline and at hospital discharge, up to 14 days after admission
  It will be evaluated using 6-min walk test according to the guideline of American Thoracic Society
Physical performance | At baseline and at hospital discharge, up to 14 days after admission
  It will evaluated using Short Physical Performance Battery.

SECONDARY OUTCOMES:
Maximum inspiratory and expiratory capacity | At baseline and at hospital discharge, up to 14 days after admission
  It will be evaluated using incentive spirometer.
Hemodynamic responses to exercise | At baseline and at hospital discharge, up to 14 days after admission
  The change in heart rate before and after exercise will be recorded
Hemodynamic responses to exercise | At baseline and at hospital discharge, up to 14 days after admission
  The change in blood pressure before and after exercise will be recorded
Hemodynamic responses to exercise | At baseline and at hospital discharge, up to 14 days after admission
  The change in oxygen saturation before and after exercise will be recorded
Subjective symptom responses to exercise | At baseline and at hospital discharge, up to 14 days after admission
  Subjective symptom responses to exercise will be evaluated by determining changes in the Modified Borg Dyspnea and Fatigue scales before and after exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University- Cerrahpasa, Cardiology Institute, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided